CLINICAL TRIAL: NCT02414789
Title: Lyme Borreliosis and Early Cutaneous Diagnostic
Acronym: DIABOLYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6084
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Erythema Migrans
Keywords: erythema migrans; Lyme; early diagnosis; skin biomarkers; proteomics diagnostic; mass spectrometry
MeSH Terms: conditions — Glossitis, Benign Migratory; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SRM / MS-MS (Experimental)
  Interventions: Procedure: Skin biopsies

INTERVENTIONS:
Procedure: Skin biopsies — Skin biopsies of patients with Lyme disease (erythema migrans) infected with Borrelia burgdorferi sensu lato will be analyzed by three diagnostic techniques : molecular technique (PCR), biological technique (culture of the bacteria) and proteomics technique (SRM/ MS-MS)

SUMMARY:
Test and evaluate a new diagnostic method (SRM-MS/MS: Selected Reaction Monitoring- Mass spectrometry) for Lyme Borreliosis on human skin biopsies. Patients included are those with the early skin manifestation (erythema migrans).

This new proteomic method will be compared to the two existing method: culture of Borrelia and PCR detection of Borrelia (DNA detection of the bacteria).

ELIGIBILITY:
Inclusion Criteria:

* Erythema migrant as criteria EUCALB or atypical form associated to tick's sting
* Patient having signed a consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Prior treatment with antibiotics
* Erythema migrans on the face
* Bleeding disorders
* Anticoagulant treatment
* Inability to give clear information (subject in an emergency situation, understanding of the topic difficulty, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Compare the sensitivity (percentage of positive tests) of the SRM / MS-MS to techniques of PCR and culture Borrelia | One year study
  percentage of positive tests with all three techniques (SRM/MS-MS ; PCR ; culture)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Centre Hospitalo-Universitaire Jean Minjoz, Besançon
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Hôpital Pasteur, Colmar
  - Hôpital E. Muller, Mulhouse
  - Hôpital Robert Debré, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Bel Air, Thionville

REFERENCES:
- [Background] Cantero P, Ehret-Sabatier L, Lenormand C, Hansmann Y, Sauleau E, Zilliox L, Westermann B, Jaulhac B, Mutter D, Barthel C, Perdu-Alloy P, Martinot M, Lipsker D, Boulanger N. Detection of Borrelia burgdorferi sensu lato by proteomics: a complementary diagnosis tool on erythema migrans biopsies. Clin Microbiol Infect. 2025 Jan;31(1):78-86. doi: 10.1016/j.cmi.2024.10.014. Epub 2024 Oct 23. PMID 39454756